CLINICAL TRIAL: NCT05476588
Title: Tobacco, Alcohol, Prescription Drug, and Illicit Substance Use- Electronic Spanish Platform
Acronym: TAPS-ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: COG Analytics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 022-114
Record Dates: First submitted 2022-07-01; First posted 2022-07-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use; Alcohol Abuse; Prescription Drug Abuse; Substance Use
MeSH Terms: conditions — Tobacco Use; Alcoholism; Substance-Related Disorders | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: randomized, two-group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administration followed by Interviewer-Administered (Active Comparator): Screening and validation of assessment tool translated into Spanish
  Interventions: Other: Screening
- Interviewer-Administered followed by Self-Administration (Active Comparator): Screening and validation of assessment tool translated into Spanish
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening and validation of assessment tool translated into Spanish

SUMMARY:
The goal of this study is to validate the TAPS-ESP as a screen and assessment that can be used in primary care for the screening and treatment of substance use.

DETAILED DESCRIPTION:
This Phase II study seeks to conduct further research to validate the TAPS-ESP as a Spanish language version of the screening and brief assessment and pave the way for its broad dissemination in the healthcare system. The investigators will use a novel application of a Type 1 hybrid effectiveness-implementation design, adapted to a screening validation study. The investigators will conduct a large-scale study to validate the TAPS-ESP against established diagnostic and biomarker metrics, replicating the design of the seminal English-language TAPS study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current patient of the clinic
* Spanish-language preferred
* Ability to read Spanish

Exclusion Criteria:

* Unable to provide informed consent
* Inability to comprehend or read Spanish
* Inability to self-administer the iPad tool due to physical limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Tobacco, Alcohol, Prescription drug, and illicit Substance Use Tool-Electronic Spanish Platform (TAPS-ESP) primary criterion validation against the modified World Mental Health Composite International Diagnostic Interview (CIDI) in Spanish | 1 year
  TAPS-ESP is a two-stage screening and assessment tool that first screens for 4 broad substance abuse categories (tobacco, alcohol, prescription drug misuse, and illicit substances), then branches to the assessment for specific risks related to an array of substances. TAPS-ESP scores will be validated against the modified World Mental Health Composite International Diagnostic Interview (CIDI) including alcohol, tobacco, and 9 substance categories. The CIDI items mapped to the diagnostic criteria for each substance will serve as the primary criterion standard for validation of the TAPS-ESP. For detecting CIDI-derived substance use disorder (SUD) diagnosis, we will examine TAPS-ESP cut-points for the 4-item screener and the assessment in detecting problem severity defined by CIDI for detecting different tiers of substance use: Problem use (1+ criteria), SUD (2+ criteria), and moderate-to-severe SUD (4-11 criteria). Detection of SUD will be the primary outcome for each substance category.

SECONDARY OUTCOMES:
Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) for concurrent and convergent validity of the TAPS Tool | 1 year
  The ASSIST was developed for the World Health Organization to screen for alcohol, tobacco, and drug use in medical care settings. For each substance, the use dimensions include lifetime use, past 3 month use, urges or cravings to use, and adverse consequences from use, as well as concerns expressed by family or friends about use (lifetime, past 3 months), failed attempts to control, cut down, or stop use (lifetime, past 3 months), and drug injection (lifetime, past 3 months). The ASSIST provides substance-specific risk scores 9 substance classes, with scores of 1-3 corresponding to low risk, 4-26 (10-26 for alcohol) to moderate risk, and 27 or higher to high risk.
Drug Abuse Screening Test (DAST-10) for concurrent and convergent validity of the TAPS Tool | 1 year
  The DAST-10 is a ten-item yes/no screen for general drug use problems (not including alcohol). Each item is worth one point, and respondents are tiered into risk categories based on score, with more intensive assessment recommended at a score of 6 or higher. It has been widely used in the substance use field, but does not distinguish between types of drugs used. A Spanish language version has been developed.
CAGE (Cut Down, Annoyed, Guilty, Eye-Opener) for concurrent and convergent validity of the TAPS | 1 year
  The CAGE is a rapid alcoholism screening test comprised of four yes/no questions (Cut Down, Annoyed, Guilty, Eye-Opener) for which ONE yes answer to any of the four items indicates DSM-IV alcohol abuse or dependence. A Spanish language version was validated in both Spain and the US, where it performed well in identifying DSM-IV alcohol abuse or dependence among Latinx primary care patients.
Alcohol Use Disorders Identification Test (AUDIT) for concurrent and convergent validity of the TAPS | 1 year
  The AUDIT is a 10-item questionnaire which covers the domains of alcohol consumption, drinking behavior, and alcohol-related problems. It was developed from a six-country World Health Organization collaborative project as a screening instrument for hazardous and harmful alcohol consumption. Responses to each of the 10 questions are scored according to a frequency rating of 0 (never) to 4 (daily), giving the entire questionnaire a possible score of 40. A score of 8 or more indicates harmful or hazardous alcohol use. A Spanish language version of the AUDIT is available.
Fagerstrom Test for Nicotine Dependence (FTND) for concurrent and convergent validity of the TAPS | 1 year
  The FTND is comprised of six questions scored on a point system, with total scoring summing between 0 and 10. Higher scores indicate heavier reliance on nicotine. The FTDN has been widely used in the tobacco field for decades. It has been found to be internally consistent and an acceptable way to measure nicotine/tobacco dependency. The FTND has been translated into Spanish and validated.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sanchez, PhD, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor Scott and White Community Care, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Two years
Access Criteria: Contact Principal Investigators

REFERENCES:
- [Derived] Gryczynski J, Sanchez K, Carswell SB, Schwartz RP. The Spanish language version of the TAPS tool: protocol for a validation and implementation study in primary care. Addict Sci Clin Pract. 2023 Nov 16;18(1):69. doi: 10.1186/s13722-023-00423-9. PMID 37974265